CLINICAL TRIAL: NCT06520488
Title: Phase IB/II Clinical Study of the Safety, Tolerability and Efficacy of HRS-4642 in Combination With Anti-tumor Agents in Subjects With Advanced Solid Tumors
Brief Title: A Study of HRS-4642 in Combination With Antineoplastic Agents in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-4642-202
Record Dates: First submitted 2024-07-22; First posted 2024-07-25 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group Part I/Part II/Part III (Experimental): Treatment group Part I: HRS-4642 combined with SHR-A1921 Treatment group Part II: HRS-4642 combined with SHR-A1904Treatment group Part II: HRS-4642 combined with AG
  Interventions: Drug: HRS-4642

INTERVENTIONS:
Drug: HRS-4642 — Treatment group Part I: HRS-4642 combined with SHR-A1921 Treatment group Part II: HRS-4642 combined with SHR-A1904 Treatment group Part II: HRS-4642 combined with AG

SUMMARY:
To evaluate the safety and preliminary efficacy of HRS-4642 in combination with antineoplastic agents in subjects with advanced solid tumors with KRAS G12D mutations, and to determine the maximum tolerated dose (MTD) and the recommended Phase II dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Age 18-75 years old (inclusive) at the time of signing the informed consent form
3. Male or female
4. ECOG score of 0 or 1
5. Expected survival ≥ 12 weeks
6. At least one measurable lesion according to RECIST v1.1 criteria

Exclusion Criteria:

1. Any other condition that, in the judgment of the investigator, may increase the risk of participating in the study, interfere with the results of the study, or be unsuitable for participation in this study
2. Presence of uncontrollable psychiatric illness and other conditions such as known alcoholism, drug or substance abuse, criminal detention, etc., that affect the completion of the study procedures
3. Known hypersensitivity to any component of HRS-4642; History of severe allergic reactions to other monoclonal antibodies/fusion protein drugs; Known history of severe hypersensitivity to antineoplastic agents in combination
4. Received other major surgery other than diagnosis or biopsy within 28 days before the first dose; Minor traumatic surgery (biopsy, laparoscopy, and drainage) within 7 days prior to the first dose; Presence of non-healing wounds (severe, non-healing, or dehiscence), untreated fractures
5. Subjects who are participating in other clinical studies or whose first dose is less than 4 weeks from the end of the previous clinical study (last dose), or who have 5 half-lives of this investigational drug, whichever is shorter
6. Use of a live attenuated vaccine within 28 days prior to the first dose of study medication, or anticipated need for a live attenuated vaccine during study treatment
7. Have a history of immunodeficiency, including a positive HIV test, other acquired or congenital immunodeficiency diseases, or a history of organ transplantation
8. Those who have active pulmonary tuberculosis infection within 1 year before enrollment, or those who have a history of active pulmonary tuberculosis infection more than 1 year ago but have not been formally treated
9. Active hepatitis B
10. Presence of clinically significant acute or chronic pancreatitis
11. Poorly controlled or severe cardiovascular and cerebrovascular diseases, arterior/venous thrombotic events within 6 months prior to study entry
12. Presence of gastrointestinal obstruction or presence of symptoms and signs of gastrointestinal obstruction within 6 months prior to the start of study treatment, but screening can be performed if surgical treatment has been performed and the obstruction has been completely resolved

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Stage 1: (IB Period):DLTs | Within 28 days of the first dose
Stage 1: (IB Period): adverse events (AEs) | Within 28 days of the first dos,About 1 year
Phase II: (Phase II):investigator-assessed ORR | Assessed every 6 weeks,About 1 year

SECONDARY OUTCOMES:
Stage 1: (IB Period):Investigator-assessed objective response rate (ORR) | Assessed every 6 weeks,About 1 year
Phase II: (Phase II):DCR | Assessed every 6 weeks,About 1 year
Phase II: (Phase II):DoR | Assessed every 6 weeks,About 1 year
Phase II: (Phase II):OS | Assessed every 6 weeks+ About 1 year
Phase II: (Phase II):PFS | Assessed every 6 weeks,About 1 year
Phase II: (Phase II):OS | Assessed approximately once every 1 month,About 1 year
Phase II: (Phase II):Incidence and severity of AEs | Assessed approximately once every 1 month,About 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided